CLINICAL TRIAL: NCT06336967
Title: A Randomized Controlled Trial of a Wellness App for First Responders, Military Personnel and Veterans
Brief Title: Testing a Wellness App for First Responders, Military Personnel and Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Nlyten Corp (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 855282
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Wellness
Keywords: first responders; veterans; soldiers; social connectedness; burnout; wellbeing
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GUIDE with incentives (Experimental): Immediate access to the GUIDE App smartphone application for 4 weeks with the opportunity to earn additional compensation, up to $100 in total, based on app engagement.
  Interventions: Behavioral: GUIDE
- GUIDE without incentives (Experimental): Immediate access to the GUIDE App for 4 weeks without the opportunity to earn additional compensation.
  Interventions: Behavioral: GUIDE
- Waitlist (No Intervention): Waitlisted with delayed access to the GUIDE App without the opportunity to earn additional compensation.

INTERVENTIONS:
Behavioral: GUIDE — The GUIDE App is a wellbeing app designed for first responders and veterans that uses small group support, a learning management system, drivers of behavior change, and an anonymous member experience safeguarded by a leader in identity and login privacy, Okta (okta.com). It includes three main features: 1) Community, 2) Wisdom, and 3) Daily Practice. The Community feature connects app users with an online community of like folks, allowing for human support, encouragement, accountability and coaching. Online communities are moderated by GUIDE employees. The Wisdom feature includes tools and interactive media for personal growth. The Daily Practice feature includes simple, daily routines to maintain mental and emotional wellness.
  Arms: GUIDE with incentives; GUIDE without incentives

SUMMARY:
The purpose of the research study is to trial a smart phone application, the GUIDE App, to better understand its impact on social connectedness, personal growth and mental health/wellness among first responders, soldiers, and veterans. The research team will also investigate workplace metrics (e.g., engagement and burnout), implementation outcomes and technical merit. The investigators plan to run a three-armed randomized waitlist pilot feasibility trial with up to 150 participants.

DETAILED DESCRIPTION:
There is an urgent need to address mental wellbeing, isolation, and burnout among first responders, military personnel and veterans. Research shows that these groups are at a greater risk for suicide, depression, and post-traumatic stress disorder (PTSD) than the general civilian population, and that their occupations make them more likely to feel isolation and burnout. Despite these risks, first responders, soldiers and veterans tend not to seek help due to stigma, time burden and other barriers to entry. The GUIDE App was designed with this population in mind. The lessons and exercises take only minutes to complete, and the group chats are anonymous, so users can share their thoughts with likeminded peers, without the stigma. In a 4-week pilot study with 16 participants from the Wilkes Barre Police Department, the GUIDE App showed promising results in promoting wellbeing, reducing anxiety and encouraging personal growth. This clinical trial builds off the pilot study. The investigators will use a three-armed randomized waitlist pilot feasibility trial with 150 participants (first responders, soldiers, and veterans) to test whether use of the GUIDE App will lead to increased social connectedness, personal growth, and mental health/wellbeing; and whether these outcomes will in turn increase work engagement and reduce burnout. The investigators will also investigate implementation outcomes (e.g., the feasibility of using the app) and technical merit (e.g., how user-friendly the app is).

ELIGIBILITY:
Inclusion Criteria:

* Law enforcement, military personnel, or veteran.
* Employed (part-time, full-time, self-employed).
* Owns compatible smartphone.
* Not paid by the GUIDE App/Nlyten Corp.
* No previous use of GUIDE App.

Exclusion Criteria:

* Not law enforcement, military personnel, or veteran.
* Not employed.
* Paid by GUIDE App/Nlyten Corp.
* Previous use of GUIDE App.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Nuske, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunphy MK, Nuske HJ. Evaluating a Mobile Health Intervention (GUIDE App) for First Responders, Military Personnel, and Veterans: Randomized Controlled Trial. J Med Internet Res. 2025 Oct 17;27:e71155. doi: 10.2196/71155. PMID 41105938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment opened on April 22, 2024 and continued through August 31, 2024. Participants were recruited through email distribution lists, GUIDE partnerships, social media posts and in-person events with the population.
Pre-assignment Details: Participants who signed the informed consent, but did not attend an introductory Zoom meeting with the clinical research coordinator, were not assigned a treatment group. Participants received app access and instructions during the introductory meeting at the meeting, which finalized their enrollment in the study.
Period: Overall Study
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Started | 39 | 37 | 39
Completed | 34 | 35 | 38
Not Completed | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Population: 2 fewer in GUIDE without incentives because of individuals who scheduled but did not attend their introductory meeting during the last week of open recruitment.
Groups:
- Total: Total of all reporting groups
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist | Total
Number analyzed (Participants) | 39 | 37 | 39 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 36 | 39 | 113
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 12 | 33
  Male | 27 | 28 | 27 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants can be counted more than once in the appropriate category.
  Participants
    White | 34 | 32 | 36 | 102
    Black or African American | 4 | 3 | 1 | 8
    American Indian/Alaska Native | 1 | 0 | 0 | 1
    Hispanic/Latino | 2 | 4 | 0 | 6
    Asian | 0 | 0 | 2 | 2
    Refused to Answer | 0 | 1 | 0 | 1
PERMA Overall Score [Mean (Standard Deviation); unit: units on a scale] — The PERMA Profiler is a validated self-report measure assessing well-being across five domains: Positive Emotion, Engagement, Relationships, Meaning, and Accomplishment. Scores range from 0 to 10, with higher scores indicating greater well-being. The PERMA Overall Score is computed by averaging the five subscale scores, each derived from three Likert-type items. Higher scores represent better well-being outcomes.
  units on a scale | 6.57 (1.43) | 7.16 (1.65) | 6.45 (1.43) | 6.72 (1.52)
Personal Wellbeing Score (PWS) [Mean (Standard Deviation); unit: score on a scale] — The Personal Wellbeing Score (PWS) is a validated self-report measure assessing subjective well-being based on the Office for National Statistics (ONS4) framework. It evaluates life satisfaction, sense of purpose, happiness, and anxiety. Scores range from 0 to 100, with higher scores indicating greater well-being. The PWS Overall Score is computed by averaging responses across four domains. Higher scores represent better well-being outcomes.
  score on a scale | 67.52 (22.52) | 77.25 (21.57) | 60.90 (24.04) | 68.41 (23.53)
WHO-5 Wellbeing [Mean (Standard Deviation); unit: score on a scale] — The WHO-5 Well-Being Index is a validated self-report measure assessing mental well-being over the past two weeks. It consists of five positively framed items, rated on a 0 to 5 Likert scale, with higher scores indicating better well-being. The total score is computed by summing item responses, then multiplying by 4 to yield a 0 to 100 scale. Scores ≤50 suggest poor well-being, and ≤28 indicate possible depression.
  score on a scale | 53.03 (21.32) | 57.30 (21.87) | 52.21 (20.66) | 54.12 (21.21)
PERMA Positive emotion [Mean (Standard Deviation); unit: units on a scale] — The PERMA Positive Emotion Score is a validated self-report measure assessing the presence of positive emotions in daily life. It is part of the PERMA Profiler, which evaluates well-being across five domains. Scores range from 0 to 10, with higher scores indicating greater positive emotional experiences. The Positive Emotion Score is computed by averaging responses to three Likert-type items. Higher scores represent better well-being outcomes.
  units on a scale | 6.07 (1.81) | 6.61 (2.09) | 5.89 (1.64) | 6.18 (1.86)
PERMA Engagement [Mean (Standard Deviation); unit: units on a scale] — The PERMA Engagement Score is a validated self-report measure assessing an individual's sense of immersion and involvement in activities. It is part of the PERMA Profiler, which evaluates well-being across five domains. Scores range from 0 to 10, with higher scores indicating greater engagement in meaningful experiences. The Engagement Score is computed by averaging responses to three Likert-type items. Higher scores represent better well-being outcomes.
  units on a scale | 6.46 (1.56) | 6.39 (1.55) | 6.72 (1.39) | 6.52 (1.50)
PERMA Relationships [Mean (Standard Deviation); unit: units on a scale] — The PERMA Relationships Score is a validated self-report measure assessing the quality and strength of social connections. It is part of the PERMA Profiler, which evaluates well-being across five domains. Scores range from 0 to 10, with higher scores indicating stronger, more supportive relationships. The Relationships Score is computed by averaging responses to three Likert-type items. Higher scores represent better well-being outcomes.
  units on a scale | 6.56 (2.07) | 7.43 (2.1) | 6.14 (1.94) | 6.70 (2.09)
PERMA Meaning [Mean (Standard Deviation); unit: units on a scale] — The PERMA Meaning Score is a validated self-report measure assessing an individual's sense of purpose and significance in life. It is part of the PERMA Profiler, which evaluates well-being across five domains. Scores range from 0 to 10, with higher scores indicating a stronger sense of meaning and purpose. The Meaning Score is computed by averaging responses to three Likert-type items. Higher scores represent better well-being outcomes.
  units on a scale | 6.91 (2.03) | 7.77 (1.95) | 6.74 (1.88) | 7.13 (1.99)
PERMA Accomplishment [Mean (Standard Deviation); unit: units on a scale] — The PERMA Accomplishment Score is a validated self-report measure assessing an individual's sense of achievement and progress toward goals. It is part of the PERMA Profiler, which evaluates well-being across five domains. Scores range from 0 to 10, with higher scores indicating greater feelings of accomplishment. The Accomplishment Score is computed by averaging responses to three Likert-type items. Higher scores represent better well-being outcomes.
  units on a scale | 6.83 (1.6) | 7.6 (1.44) | 6.74 (1.6) | 7.05 (1.59)
PERMA Happiness [Mean (Standard Deviation); unit: units on a scale] — The PERMA Happiness Score is a validated self-report measure assessing an individual's overall sense of joy and life satisfaction. It is part of the PERMA Profiler, which evaluates well-being across five domains. Scores range from 0 to 10, with higher scores indicating greater happiness. The Happiness Score is computed by averaging responses to three Likert-type items. Higher scores represent better well-being outcomes.
  units on a scale | 6.64 (1.91) | 6.89 (1.90) | 6.31 (1.81) | 6.61 (1.87)
PERMA Health [Mean (Standard Deviation); unit: units on a scale] — The PERMA Health Score is a validated self-report measure assessing an individual's subjective sense of physical health and vitality. It is part of the PERMA Profiler, which evaluates well-being across multiple domains. Scores range from 0 to 10, with higher scores indicating better perceived health. The Health Score is computed by averaging responses to three Likert-type items. Higher scores represent better well-being outcomes.
  units on a scale | 6.01 (1.69) | 6.80 (1.83) | 5.54 (1.77) | 6.10 (1.82)
PERMA Negative emotion [Mean (Standard Deviation); unit: units on a scale] — The PERMA Negative Emotion Score is a validated self-report measure assessing the presence of distressing emotions such as sadness, anxiety, and anger. It is part of the PERMA Profiler, which evaluates well-being across multiple domains. Scores range from 0 to 10, with higher scores indicating greater negative emotional experiences. The Negative Emotion Score is computed by averaging responses to three Likert-type items. Lower scores represent better well-being outcomes.
  units on a scale | 4.45 (2.18) | 3.81 (1.93) | 4.22 (1.74) | 4.17 (1.96)
PERMA Loneliness [Mean (Standard Deviation); unit: units on a scale] — The PERMA Loneliness Score is a validated self-report measure assessing an individual's sense of social isolation and lack of connection. It is part of the PERMA Profiler, which evaluates well-being across multiple domains. Scores range from 0 to 10, with higher scores indicating greater feelings of loneliness. The Loneliness Score is computed by averaging responses to three Likert-type items. Lower scores represent better well-being outcomes.
  units on a scale | 3.69 (2.99) | 3.57 (2.77) | 5.13 (3.10) | 4.14 (3.02)
DERS-SF [Mean (Standard Deviation); unit: units on a scale] — The Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) is a validated self-report measure assessing emotion regulation difficulties across six domains: nonacceptance of emotions, goal-directed behavior, impulse control, emotional awareness, access to regulation strategies, and emotional clarity. Scores range from 18 to 90, with higher scores indicating greater difficulties in emotion regulation. The DERS-SF Total Score is computed by summing responses across all items. Lower scores represent better emotion regulation outcomes.
  units on a scale | 36.54 (12.59) | 31.19 (10.17) | 39.00 (12.46) | 35.65 (12.16)
Anxiety (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder 7-item (GAD-7) is a validated self-report measure assessing anxiety symptom severity over the past two weeks. It consists of seven items, rated on a 0 to 3 Likert scale, with higher scores indicating greater anxiety severity. The total score is computed by summing item responses, yielding a 0 to 21 scale. Scores of 5, 10, and 15 indicate mild, moderate, and severe anxiety, respectively.
  units on a scale | 13.36 (5.73) | 11.00 (4.34) | 13.54 (4.32) | 12.66 (4.95)
Depression (PHQ-8) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-8 (PHQ-8) is a validated self-report measure assessing depressive symptom severity over the past two weeks. It consists of eight items, rated on a 0 to 3 Likert scale, with higher scores indicating greater depression severity. The total score is computed by summing item responses, yielding a 0 to 24 scale. Scores of 5, 10, 15, and 20 indicate mild, moderate, moderately severe, and severe depression, respectively.
  units on a scale | 7.36 (5.15) | 5.14 (5.05) | 7.51 (5.19) | 6.70 (5.20)

OUTCOME MEASURES:

1. Primary Outcome: PERMA-Profiler Overall Wellbeing Score
Description: The PERMA-Profiler is designed to measure the general wellbeing of adults; specifically this questionnaire measures positive and negative emotions, engagement, relationships, meaning, accomplishment, and health. Participants respond to 23 items on an 11-point Likert scale, from 0 to 10. Scores are calculated as the average of the items comprising each factor. Lower scores indicate lower flourishing, and higher scores indicate higher flourishing.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analyzed data for all participants who completed the post-trial assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
score on a scale | 6.99 (1.47) | 7.46 (1.62) | 6.49 (1.58)

2. Primary Outcome: Patient Health Questionnaire for Depression Symptoms (PHQ-8)
Description: The PHQ-8 is a self-reported measure of depressive symptoms composed of 8 Likert type items with a response scale ranging from 0 (Not at all) to 3 (Nearly every day), that refer to the presence of that symptom during the previous 2 weeks. Each item corresponds to the first 8 symptoms of the 4th edition of the DSM-IV diagnostic criteria for major depressive disorder. The PHQ-8 final score is obtained by adding the score for each of the items, ranging from 0 to 24 (higher scores corresponding to higher levels of depression).
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed their post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 5.15 (3.509) | 3.86 (3.844) | 6.29 (4.667)

3. Primary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: GAD-7 consists of seven items measuring worry and anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity. Scores above 10 are considered to be in the clinical range. The GAD-7 has shown good reliability and construct validity.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analyzed for all participants who completed a post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 12.53 (5.089) | 10.34 (3.235) | 13.42 (4.665)

4. Primary Outcome: WHO Well-being Index (WHO-5)
Description: The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. The WHO-5 consists of five statements, which respondents rate according to the scale below (in relation to the past two weeks).
  All of the time = 5 Most of the time = 4 More than half of the time = 3 Less than half of the time = 2 Some of the time = 1 At no time = 0.
  The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed their post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 57.41 (19.394) | 65.71 (19.239) | 52.95 (21.838)

5. Primary Outcome: Personal Wellbeing Score (PWS)
Description: The Personal Wellbeing Score (PWS) is based on the Office of National Statistics (ONS) four subjective well-being questions (ONS4) and thresholds. It evaluates life satisfaction, sense of purpose, happiness, and anxiety. Each PWS item is scored as follows: Disagree=0, Neutral=1, Agree=2 and Strongly Agree=3. Summary scores are calculated by aggregating all items and transforming to a scale of 0 to 100, with higher scores indicating greater well-being.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 73.04 (24.11) | 77.62 (18.72) | 62.28 (22.24)

6. Primary Outcome: Difficulties in Emotion Regulation Scale Short Form (DERS-SF)
Description: The Difficulties in Emotion Regulation Scale Short Form (DERS-SF) is an 18-item measure used to identify emotional regulation issues in adults. The measure uses 6 subscales to measure 4 dimensions of emotional regulation: awareness; acceptance; the ability to engage in goal-directed behavior and refrain from impulsive behavior when experiencing negative emotions; and access to emotion regulation strategies perceived as effective. Respondents indicate how often each statement applies to them on a 5 point scale, where 1=Almost Never (0-10%), 2=Sometimes (11-35%), About Half of the Time (36-65%), Most of the Time (66-90%), Almost Always (91-100%). Scores range from 18 to 90, with higher scores indicating greater difficulties in emotion regulation. The DERS-SF Total Score is computed by summing responses across all items. Lower scores represent better emotion regulation outcomes.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed a post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 32.82 (9.974) | 32.06 (9.825) | 36.89 (11.795)

7. Secondary Outcome: Positive Emotion (Positive Emotion Subscale of the PERMA-Profiler)
Description: The PERMA-Profiler is a 23-item measure that assesses wellbeing across five domains (positive emotion, engagement, relationships, meaning, accomplishment). The instrument was constructed so that each domain can be defined and measured as separate but correlated constructs. This study will use the Positive Emotion subscale of the PERMA. This subscale includes 3 items on an 11-point Likert scale, from 0 to 10. Scores are calculated as an average of these items, with lower scores indicating less positive emotion and high scores indicating more positive emotion.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 6.65 (1.65) | 7.20 (1.89) | 5.96 (1.87)

8. Secondary Outcome: Social Connectedness (Engagement Subscale of PERMA-Profiler)
Description: The PERMA-Profiler is a 23-item measure that assesses wellbeing across five domains (positive emotion, engagement, relationships, meaning, accomplishment). The instrument was constructed so that each domain can be defined and measured as separate but correlated constructs. This study will use the Engagement and Relationship subscales of the PERMA. These subscales include 3 items each, ranked on an 11-point Likert scale, from 0 to 10. Scores are calculated as an average of these items for each subscale, with lower scores indicating less flourishing in respect to engagement/relationships and high scores indicating better engagement/relationships.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed a post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 6.66 (1.43) | 6.70 (1.77) | 6.68 (1.53)

9. Secondary Outcome: Social Connectedness (Relationship Subscale of PERMA-Profiler)
Description: as for outcome 8
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed a post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 7.03 (2.03) | 7.81 (2.03) | 6.14 (1.93)

10. Secondary Outcome: Personal Growth (Meaning Subscale of the PERMA-Profiler)
Description: The PERMA-Profiler is a 23-item measure that assesses wellbeing across five domains (positive emotion, engagement, relationships, meaning, accomplishment). The instrument was constructed so that each domain can be defined and measured as separate but correlated constructs. This study will use the Meaning and Accomplishment subscales of the PERMA. These subscales include 3 items each, ranked on an 11-point Likert scale, from 0 to 10. Scores are calculated as an average of these items for each subscale, with lower scores indicating less flourishing in respect to meaning/accomplishment and high scores indicating more meaning/accomplishment.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes participants who completed their post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 7.33 (1.92) | 7.86 (1.88) | 6.74 (2.10)

11. Secondary Outcome: Personal Growth (Accomplishment Subscale of the PERMA-Profiler)
Description: as for outcome 10
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes participants who completed their post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 7.29 (1.46) | 7.74 (1.49) | 6.95 (1.65)

12. Secondary Outcome: Utrecht Work Engagement Scale (UWES-17)
Description: The Utrecht Work Engagement Scale-17 assesses work engagement, or a positive, fulfilling, work-related state of mind characterized by vigor, dedication, and absorption. It is intended to measure the 'opposite' of burnout in both university students and employees. Items were developed to reflect three underlying dimensions: "Vigor" (VI); "Dedication" (DE), and "Absorption" (AB). The subscales were found to be internally consistent but relatively strongly correlated. Items are scored along a 6-point Likert-type scale (0 = Never to 6 = Always or Every day). Scores are calculated by summing item scores. The total score ranges from 0 to 102 points. A higher score indicates greater worker engagement.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 61.74 (17.647) | 62.49 (14.496) | 58.61 (16.668)

13. Secondary Outcome: Maslach Burnout Inventory (MBI) - Emotional Exhaustion
Description: The Maslach Burnout Inventory - Emotional Exhaustion (MBI-EE) is a validated self-report measure assessing feelings of emotional depletion and fatigue due to work-related stress. It is part of the Maslach Burnout Inventory (MBI), which evaluates burnout across three domains. Scores range from 0 to 54, with higher scores indicating greater emotional exhaustion. The Emotional Exhaustion Score is computed by summing responses to nine Likert-type items. Lower scores represent better well-being outcomes.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 21.24 (12.015) | 19.06 (10.287) | 19.97 (11.507)

14. Secondary Outcome: Maslach Burnout Inventory (MBI) - Personal Accomplishment
Description: The Maslach Burnout Inventory - Personal Accomplishment (MBI-PA) is a validated self-report measure assessing feelings of competence and achievement in one's work. It is part of the Maslach Burnout Inventory (MBI), which evaluates burnout across three domains. Scores range from 0 to 48, with higher scores indicating greater personal accomplishment and lower scores suggesting burnout-related inefficacy. The Personal Accomplishment Score is computed by summing responses to eight Likert-type items.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 31.38 (8.739) | 32.00 (6.924) | 30.42 (7.866)

15. Secondary Outcome: Maslach Burnout Inventory (MBI) - Depersonalization
Description: The Maslach Burnout Inventory - Depersonalization (MBI-DP) is a validated self-report measure assessing feelings of detachment and impersonal responses toward others in a work setting. It is part of the Maslach Burnout Inventory (MBI), which evaluates burnout across three domains. Scores range from 0 to 30, with higher scores indicating greater depersonalization and emotional distancing. The Depersonalization Score is computed by summing responses to five Likert-type items. Lower scores represent better well-being outcomes.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Analysis includes all participants who completed post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
units on a scale | 8.79 (6.285) | 8.86 (6.335) | 9.13 (6.156)

16. Secondary Outcome: Number of Participants Still Employed
Description: Whether the participant still has their job at the end of the 4-week trial period.
Time Frame: assessed at Baseline and post-trial (over 4 weeks), post-trial (week 4) reported
Population: Only included participants who completed their post-trial assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives | Waitlist
Number analyzed (Participants) | 34 | 35 | 38
Participants | 34 | 35 | 38

17. Secondary Outcome: Feasibility of Intervention Measure (FIM)
Description: The Feasibility of Intervention Measure (FIM) is used to measure the feasibility of an intervention. The scale consists of 4 items rated on a 5-point Likert Scale from 1 ("Completely disagree") to 5 ("Completely agree"). The score consists of the average of the items, ranging from 1 to 5, with higher scores indicating greater feasibility of the intervention.
Time Frame: assessed at post-trial (4 weeks)
Population: Included participants from two groups that used GUIDE during the trial, only if they completed their post-trial assessment survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives
Number analyzed (Participants) | 34 | 35
units on a scale | 3.941176471 (0.89200749) | 4.078571429 (0.638159776)

18. Secondary Outcome: Acceptability of Intervention Measure (AIM)
Description: The Acceptability of Intervention Measure (AIM) is used to measure the acceptability of an intervention. The scale consists of 4 items rated on a 5-point Likert Scale from 1 ("Completely disagree") to 5 ("Completely agree"). The score consists of the average of the items, ranging from 1 to 5, with higher scores indicating greater acceptability of the intervention.
Time Frame: 4 weeks post-trial
Population: Includes: 1) participants from groups who used GUIDE during the trial, 2) participants who completed their post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives
Number analyzed (Participants) | 34 | 35
units on a scale | 3.757352941 (1.00469597) | 3.878571429 (0.777371676)

19. Secondary Outcome: Intervention Appropriateness Measure (IAM)
Description: The Intervention Appropriateness Measure (IAM) is used to measure the appropriateness of an intervention. The scale consists of 4 items rated on a 5-point Likert Scale from 1 ("Completely disagree") to 5 ("Completely agree"). The score consists of the average of the items, ranging from 1 to 5, with higher scores indicating greater appropriateness of the intervention.
Time Frame: 4 weeks post-trial
Population: Includes participants who: 1) assigned to a group that used GUIDE during the trial, 2) completed post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives
Number analyzed (Participants) | 34 | 35
units on a scale | 3.933823529 (0.817212612) | 4.085714286 (0.69118094)

20. Secondary Outcome: System Usability Scale (SUS)
Description: The System Usability Scale (SUS) measures perceptions of usability of a given system, in this case, the GUIDE App. The scale consists of 10 items, each rated on a 5-point Likert Scale from 1 ("Strongly disagree") to 5 ("Strongly agree"). Responses are transformed to get a total range of possible values from 0-100, with higher scores indicating higher perceptions of usability. Typically, a score above 68 is regarded as a good score.
Time Frame: 4 weeks post-trial
Population: Analysis includes participants who: 1) used GUIDE for the trial period, 2) completed their post-trial assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GUIDE With Incentives | GUIDE Without Incentives
Number analyzed (Participants) | 34 | 35
units on a scale | 70.07352941 (19.0442596) | 71.14285714 (18.85843992)

ADVERSE EVENTS:
Time Frame: 5 months 10 days (22 April 2024-01 October 2024)
Description: We collected information about adverse events during virtual post-trial meetings with participants who used GUIDE.
Groups:
- Intervention: GUIDE With Incentives: Immediate access to the GUIDE App smartphone application for 4 weeks with the opportunity to earn additional compensation, up to $100 in total, based on app engagement.
  GUIDE: The GUIDE App is a wellbeing app designed for first responders and veterans that uses small group support, a learning management system, drivers of behavior change, and an anonymous member experience safeguarded by a leader in identity and login privacy, Okta (okta.com). It includes three main features: 1) Community, 2) Wisdom, and 3) Daily Practice. The Community feature connects app users with an online community of like folks, allowing for human support, encouragement, accountability and coaching. Online communities are moderated by GUIDE employees. The Wisdom feature includes tools and interactive media for personal growth. The Daily Practice feature includes simple, daily routines to maintain mental and emotional wellness.
- Intervention: GUIDE Without Incentives: Immediate access to the GUIDE App for 4 weeks without the opportunity to earn additional compensation.
  GUIDE: The GUIDE App is a wellbeing app designed for first responders and veterans that uses small group support, a learning management system, drivers of behavior change, and an anonymous member experience safeguarded by a leader in identity and login privacy, Okta (okta.com). It includes three main features: 1) Community, 2) Wisdom, and 3) Daily Practice. The Community feature connects app users with an online community of like folks, allowing for human support, encouragement, accountability and coaching. Online communities are moderated by GUIDE employees. The Wisdom feature includes tools and interactive media for personal growth. The Daily Practice feature includes simple, daily routines to maintain mental and emotional wellness.
- Waitlist: No Intervention: Waitlisted with delayed access to the GUIDE App without the opportunity to earn additional compensation.
Arm/Group | Intervention: GUIDE With Incentives | Intervention: GUIDE Without Incentives | Waitlist: No Intervention
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/37 | 0/39

LIMITATIONS AND CAVEATS:
1) we relied exclusively on subjective self-report data in the trial. 2) our sample includes only those motivated enough to voluntarily participate in a clinical trial to test a mental health and wellness app, which may not be representative of this population. 3) participants were higher than average in anxiety and depression symptoms as compared to other studies of first responders and military, indicating that generalizability may be difficult. 4) short follow-up period. 5) not blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT06336967/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT06336967/ICF_001.pdf